CLINICAL TRIAL: NCT00140218
Title: Futility Study of R(+) Pramipexole in Early Amyotrophic Lateral Sclerosis
Brief Title: R(+) Pramipexole in Early Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bennett, James P., Jr., M.D., Ph.D. (Individual)
Collaborators: University of Pittsburgh (Other)
Responsible Party: James P. Bennett Jr. M.D. Ph.D. Sponsor, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11736
Expanded Access: Available
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2008-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; pramipexole; oxidative stress; neuroprotection
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: R(+) pramipexole dihydrochloride monohydrate — 10 mg tid oral

SUMMARY:
The hypothesis of this study is that treatment with R(+) pramipexole at 30 mg/day will alter the slope of decline in ALS functional rating scale over the course of 6 months. ALS patients at an early stage of disease will be observed for 3 months after enrollment and then treated with drug for 6 months.

DETAILED DESCRIPTION:
This is a futility design Phase II study using ALS-FRSr as the primary variable to monitor progression of disease in patients with early ALS. The drug to be tested is R(+) pramipexole, an antioxidant that concentrates into brain and mitochondria. R(+)PPX will be administered at 30 mg/day over 6 months, following a 3 month lead-in period without drug therapy. For purposes of this study, futility is defined as failure to decrease the slope of ALS-FRSr decline by less than 40%.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of ALS FVC>60% of predicted not being ventilated no difficulty swallowing ambulatory (can use assistance devices)

Exclusion Criteria:

* ALS duration >3 years advanced ALS with survival predicted <6 months dementia (MMSE<22) prior exposure to R(+) pramipexole orthostatic hypotension >30 mmHg history of psychosis or hallucinations abnormal baseline safety lab values

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2007-01 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
ALS-FRSr score taken each month for 3 months during lead-in and for 6 months during treatment | -3 -2 -1 0 1 2 3 4 5 6 months

SECONDARY OUTCOMES:
FVC taken each month | -3 -2 -1 0 1 2 3 4 5 6 months
hand dynamometry taken each month | -3 -2 -1 0 1 2 3 4 5 6

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence H Phillips, M.D., Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - David Lacomis MD, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia